CLINICAL TRIAL: NCT00455078
Title: The Role of Reflux in Innate Immunity Activation After Lung Transplantation.
Brief Title: GI Reflux in Lung Transplant and Its Relationship to Chronic Rejection
Acronym: LTXGERD
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 15272A
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastric reflux; Lung transplant; chronic rejection; Gastric reflux in lung transplant as it relates to chronic rejection
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: esophagogastroduodenoscopy — EGD will be done pretransplant then again before 18mos post transplant.
Other: Standard GER questionnaire (RDQ) — RDQ questionnaire will be done pretransplant then again before 18mos post transplant.
Procedure: Scintigraphic evaluation of solid gastric emptying — Scintigraphic evaluation of solid gastric emptying will be done pretransplant then again before 18mos post transplant.
Procedure: Twenty-four hour ambulatory pH testing — Twenty-four hour ambulatory pH testing will be done pretransplant then again before 18mos post transplant.
Procedure: Esophageal manometry testing — Esophageal manometry testing will be done pretransplant then again before 18mos post transplant.

SUMMARY:
Recent data has suggested that GER (gastric reflux) may worsen after lung transplantation and potentially increase the risk of chronic rejection (CR) after lung transplantation.

The purpose of this study is to look at how often GER occurs in the lung transplant population and examine how GER may change the immune system and cause CR. In this way, we would be able to better identify patients that may benefit from anti-reflux procedures.

DETAILED DESCRIPTION:
Part of standard pre-transplant work up includes a gastrointestinal (GI) work-up to check for GER. The following procedures will be done pre-transplant.

1. Standard GER questionnaire (RDQ): This is a 12 item questionnaire. This questionnaire will ask questions about any reflux symptoms present.
2. Esophagogastroduodenoscopy (EGD): This test will determine evidence of esophageal reflux and presence of a hiatal hernia.
3. Scintigraphic evaluation of solid gastric emptying: This measures the speed with which food empties from the stomach and enters the small intestine.
4. Twenty-four hour ambulatory pH testing: The ambulatory 24-hour pH monitoring test will monitor the acid in the esophagus during a 24-hour period.
5. Esophageal manometry testing: This procedure is done to evaluate the cause of reflux of stomach acid and contents back into the esophagus, and to determine the cause of problems with swallowing food.

These procedures will be done again at 3 to 6 months post transplant. The results of the EGD, scintigraphic evaluation, answers of RDQ, pH testing, esophageal manometry and bronchoscopy will be collected as well as spirometries and any episodes of rejection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing pre-lung transplant evaluations at the University of Chicago Hospital
* Patients who are capable of becoming pregnant must have a negative pregnancy test prior to consent.
* All patients must be able to give written informed consent.

Exclusion Criteria:

* Pre-transplant patients in whom study procedures are contraindicated or patients who are unable to complete all the study procedures.
* Patients who are unable to give consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone pretransplant evaluation and are on the waiting list or subjects transplanted < 18mos.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta M. Bhorade, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States